CLINICAL TRIAL: NCT00850577
Title: A Randomized Double-Blinded Phase II Study of Carboplatin/Paclitaxel/CT-322 Versus Carboplatin/Paclitaxel/Bevacizumab as First-Line Treatment for Recurrent or Advanced Non-Small Cell Lung Cancer With Non-Squamous Histology
Brief Title: Ph II of a Novel Anti-angiogenic Agent in Combination With Chemotherapy for the Treatment of Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA196-005; EUDRACT# 2008-007768-41
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; CT-322; Bevacizumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel/Carboplatin/CT-322 (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: CT-322
- Paclitaxel/Carboplatin/Bevacizumab/Placebo (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab; Drug: Bevacizumab placebo (ie saline solution)

INTERVENTIONS:
Drug: Paclitaxel — Solution, IV, 200 mg/m2, Q21days, 6 cycles
  Other Names: Taxol
Drug: Carboplatin — Solution, IV, AUC=6, Q21days, 6 cycles
  Other Names: Paraplatin
Drug: CT-322 — Solution, IV, 2 mg/kg, Q7days, Until PD
  Other Names: BMS-844203
  Arms: Paclitaxel/Carboplatin/CT-322
Drug: Bevacizumab — Solution, IV, 15 mg/kg, Q21days, Until PD
  Other Names: Avastin
  Arms: Paclitaxel/Carboplatin/Bevacizumab/Placebo
Drug: Bevacizumab placebo (ie saline solution) — Solution, IV, 0 mg/kg, On days 8 and 15 of a 3-weekly cycle, Until PD
  Other Names: Saline solution
  Arms: Paclitaxel/Carboplatin/Bevacizumab/Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of CT-322 comparative to bevacizumab, both in combination with carboplatin and paclitaxel in the treatment of chemonaive subjects with recurrent or advanced non-squamous NSCLC

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* ECOG Performance Status (PS) <=1
* Histologically or cytologically confirmed, stage IIIB (malignant pleural effusion), stage IV or recurrent NSCLC
* Measurable disease by RECIST guidelines

Exclusion Criteria:

* Evidence of predominantly squamous-cell histology
* Known CNS metastases
* Any prior antineoplastic systemic regimens for NSCLC
* Excessive risk of bleeding (including use of therapeutic anticoagulation) and history of thrombotic or embolic cerebrovascular accident
* Gross hemoptysis (≥1/2 tsp of red blood)
* Uncontrolled hypertension
* Clinically significant cardiovascular disease
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Serious non-healing wound, active peptic ulcer, non-healing bone fracture, or bleeding skin metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Progression free survival based on tumor assessments (CT scans/MRI) | every 6 weeks until documented progressive disease , death or initiation of subsequent therapy for NSCLC

SECONDARY OUTCOMES:
Overall survival (OS) between 2 arms | every 12 weeks
Objective tumor response rate (ORR) between 2 arms | every 6 weeks
Safety in the CT-322 plus carboplatin and paclitaxel arm | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (51):
- United States (20):
  - Acrc/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Sharp Clinical Oncology Research, San Diego, California
  - Cancer Institute Of Florida, Orlando, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Clintell, Inc., Skokie, Illinois
  - Cancer Center Of Kansas, Wichita, Kansas
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Annapolis Oncology Center, Annapolis, Maryland
  - Meritus Center For Clinical Research, Hagerstown, Maryland
  - North Mississippi Hematology And Oncology Associates, Ltd, Tupelo, Mississippi
  - Piedmont Hematology Oncology Associates, Pllc, Winston-Salem, North Carolina
  - North Canton Medical Clinic Center, Canton, Ohio
  - Kaiser Permanente Oncology/Hematology, Portland, Oregon
  - Guthrie Clinic, Ltd, Sayre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Charleston Hematology Oncology Associates, Pa, Charleston, South Carolina
  - Cancer Center At Cookeville Regional Medical Center, Cookeville, Tennessee
  - University Of Tennessee Cancer Institute, Memphis, Tennessee
  - Blue Ridge Cancer Care, Christiansburg, Virginia
  - Providence Western Washington Oncology, Lacey, Washington
- Brazil (6):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Rio de Janeiro, Rio de Janeiro
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, São Paulo, São Paulo
- France (5):
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Toulouse
  - Local Institution, Tours
- Italy (5):
  - Local Institution, Meldola (Fc)
  - Local Institution, Ravenna
  - Local Institution, Rimini
  - Local Institution, Roma
  - Local Institution, Terni
- Poland (6):
  - Local Institution, Bialystok
  - Local Institution, Gdansk
  - Local Institution, Otwock
  - Local Institution, Poznan
  - Local Institution, Szczecin
  - Local Institution, Warsaw
- Russia (3):
  - Local Institution, Chelyabinsk
  - Local institution, Ivanovo
  - Local Institution, Moscow
- South Africa (4):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Rondebosch, Western Cape
- United Kingdom (2):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Leeds, West Yorkshire

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx